CLINICAL TRIAL: NCT04736043
Title: Development of a Prediction Platform for Adjuvant Treatment and Prognosis in Pancreatic Cancer Using Ex Vivo Analysis of Organoid Culture
Brief Title: Development of a Prediction Platform for Adjuvant Treatment and Prognosis in Resected Pancreatic Cancer Using Organoid
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, JooKyung Park, Associate Professor, Samsung Medical Center
Other Study IDs: 2020-12-106-001
Record Dates: First submitted 2021-01-26; First posted 2021-02-03 (Actual); Last update posted 2021-02-03 (Actual); Status verified 2021-01

CONDITIONS: Pancreatic Cancer Resectable

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with resected pancreatic cancer who require adjuvant chemotherapy
  Interventions: Other: Organoid

INTERVENTIONS:
Other: Organoid — The investigators create organoid from the pancreatic cancer tissue obtained via EUS-FNA and EUS-FNB within the pancreatic cancer diagnostic process. And also the investigators create organoid from the pancreatic cancer tissue obtained after surgery as part of the pancreatic cancer treatment process. Check for the reactivity to anti-cancer drugs through cell viability assay after treating with various anti-cancer drugs, such as anti-cancer drugs used as adjuvant chemotherapy for pancreatic cancer to the organoid. Also, perform genomic analysis on each organoid, and then check if there are any unique genomic mutations for each organoid. By recognizing the relationship between the unique genomic mutations and reactivity to the anti-cancer drug within pancreatic cancer patients eligible for surgery, the investigators aim to strategize appropriate adjuvant chemotherapy after surgery, thus developing a platform to predict the outcomes of each patient.

SUMMARY:
The investigators create organoid from the pancreatic cancer tissue obtained via EUS-FNA and EUS-FNB within the pancreatic cancer diagnostic process. And also the investigators create organoid from the pancreatic cancer tissue obtained after surgery as part of the pancreatic cancer treatment process. Check for the reactivity to anti-cancer drugs through cell viability assay after treating with various anti-cancer drugs, such as anti-cancer drugs used as adjuvant chemotherapy for pancreatic cancer to the organoid. Also, perform genomic analysis on each organoid, and then check if there are any unique genomic mutations for each organoid. By recognizing the relationship between the unique genomic mutations and reactivity to the anti-cancer drug within pancreatic cancer patients eligible for surgery, the investigators aim to strategize appropriate adjuvant chemotherapy after surgery, thus developing a platform to predict the outcomes of each patient.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years old or older
2. Newly discovered pancreatic cancer and not a relapse
3. Diagnosed with pancreatic cancer via EUS-FNA, EUS-FNB before surgery
4. Patients who can undergo surgery for pancreatic cancer
5. Diagnosed with pancreatic cancer from the final tissue pathology diagnosis after surgery
6. who is in need of adjuvant chemotherapy after surgery
7. Able to make decisions for oneself for participation
8. Has obtained voluntary consent in written form (if 70 years of age or older, receive consent from the guardian as well)

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A patient who is in need of adjuvant chemotherapy after surgery, having been diagnosed with pancreatic cancer via EUS-FNA and EUS-FNB at Samsung Medical Center
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2021-01-31 (Estimated); Primary Completion 2025-01-07 (Estimated); Study Completion 2026-01-07 (Estimated)

PRIMARY OUTCOMES:
Overall survival rate | From date of initiation of adjuvant chemotherapy after surgery until the date of death from any cause, assessed up to 36 months
  The percentage of people in a group who are still alive for a certain period of time after they were started adjuvant chemotherapy for pancreatic cancer

CONTACTS AND LOCATIONS:
Locations (1):
- Samsung Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ito Y, Inoue E, Matsui Y, Kobuchi S, Moyama C, Amagase K, Yoshimura M, Ikehara Y, Nakata S, Nakanishi H. Cytology-based Detection of Circulating Tumour Cells in Human Pancreatic Cancer Xenograft Models With KRAS Mutation. Anticancer Res. 2020 Dec;40(12):6781-6789. doi: 10.21873/anticanres.14701. PMID 33288571
- [Background] Huang L, Bockorny B, Paul I, Akshinthala D, Frappart PO, Gandarilla O, Bose A, Sanchez-Gonzalez V, Rouse EE, Lehoux SD, Pandell N, Lim CM, Clohessy JG, Grossman J, Gonzalez R, Del Pino SP, Daaboul G, Sawhney MS, Freedman SD, Kleger A, Cummings RD, Emili A, Muthuswamy LB, Hidalgo M, Muthuswamy SK. PDX-derived organoids model in vivo drug response and secrete biomarkers. JCI Insight. 2020 Nov 5;5(21):e135544. doi: 10.1172/jci.insight.135544. PMID 32990680
- [Background] Ni XG, Bai XF, Mao YL, Shao YF, Wu JX, Shan Y, Wang CF, Wang J, Tian YT, Liu Q, Xu DK, Zhao P. The clinical value of serum CEA, CA19-9, and CA242 in the diagnosis and prognosis of pancreatic cancer. Eur J Surg Oncol. 2005 Mar;31(2):164-9. doi: 10.1016/j.ejso.2004.09.007. PMID 15698733
- [Background] Brody JR, Witkiewicz AK, Yeo CJ. The past, present, and future of biomarkers: a need for molecular beacons for the clinical management of pancreatic cancer. Adv Surg. 2011;45:301-21. doi: 10.1016/j.yasu.2011.04.002. No abstract available. PMID 21954696
- [Background] Leary RJ, Kinde I, Diehl F, Schmidt K, Clouser C, Duncan C, Antipova A, Lee C, McKernan K, De La Vega FM, Kinzler KW, Vogelstein B, Diaz LA Jr, Velculescu VE. Development of personalized tumor biomarkers using massively parallel sequencing. Sci Transl Med. 2010 Feb 24;2(20):20ra14. doi: 10.1126/scitranslmed.3000702. PMID 20371490
- [Background] McKernan KJ, Peckham HE, Costa GL, McLaughlin SF, Fu Y, Tsung EF, Clouser CR, Duncan C, Ichikawa JK, Lee CC, Zhang Z, Ranade SS, Dimalanta ET, Hyland FC, Sokolsky TD, Zhang L, Sheridan A, Fu H, Hendrickson CL, Li B, Kotler L, Stuart JR, Malek JA, Manning JM, Antipova AA, Perez DS, Moore MP, Hayashibara KC, Lyons MR, Beaudoin RE, Coleman BE, Laptewicz MW, Sannicandro AE, Rhodes MD, Gottimukkala RK, Yang S, Bafna V, Bashir A, MacBride A, Alkan C, Kidd JM, Eichler EE, Reese MG, De La Vega FM, Blanchard AP. Sequence and structural variation in a human genome uncovered by short-read, massively parallel ligation sequencing using two-base encoding. Genome Res. 2009 Sep;19(9):1527-41. doi: 10.1101/gr.091868.109. Epub 2009 Jun 22. PMID 19546169
- [Background] Ware JS, Roberts AM, Cook SA. Next generation sequencing for clinical diagnostics and personalised medicine: implications for the next generation cardiologist. Heart. 2012 Feb;98(4):276-81. doi: 10.1136/heartjnl-2011-300742. Epub 2011 Nov 29. PMID 22128206
- [Background] Kiyonami R, Schoen A, Prakash A, Peterman S, Zabrouskov V, Picotti P, Aebersold R, Huhmer A, Domon B. Increased selectivity, analytical precision, and throughput in targeted proteomics. Mol Cell Proteomics. 2011 Feb;10(2):M110.002931. doi: 10.1074/mcp.M110.002931. Epub 2010 Jul 27. PMID 20664071
- [Background] Campbell PJ, Yachida S, Mudie LJ, Stephens PJ, Pleasance ED, Stebbings LA, Morsberger LA, Latimer C, McLaren S, Lin ML, McBride DJ, Varela I, Nik-Zainal SA, Leroy C, Jia M, Menzies A, Butler AP, Teague JW, Griffin CA, Burton J, Swerdlow H, Quail MA, Stratton MR, Iacobuzio-Donahue C, Futreal PA. The patterns and dynamics of genomic instability in metastatic pancreatic cancer. Nature. 2010 Oct 28;467(7319):1109-13. doi: 10.1038/nature09460. PMID 20981101